CLINICAL TRIAL: NCT03428373
Title: Rivaroxaban for Improvement of Thromboembolism Outcomes in Patients With Multiple Myeloma on Lenalidomide-based Therapy: RithMM Trial
Brief Title: Rivaroxaban or Aspirin As Thromboprophylaxis in Multiple Myeloma
Acronym: RithMM
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Ottawa Hospital (Other); Dalhousie University (Other); Niagara Health System (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 110804
Record Dates: First submitted 2016-09-21; First posted 2018-02-09 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma Progression; Multiple Myeloma Stage II; Multiple Myeloma Stage I; Multiple Myeloma With Failed Remission; Multiple Myeloma Stage III
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Len-Dex+Rivaroxaban (Experimental): Patients with MM will receive Len-Dex combination and Rivaroxaban (10 mg) daily
  Interventions: Drug: Rivaroxaban
- Len-Dex+ASA (Active Comparator): Patients MM will receive Len-Dex combination and ASA 81 mg daily
  Interventions: Drug: ASA

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 10mg daily
  Other Names: Xarelto
  Arms: Len-Dex+Rivaroxaban
Drug: ASA — ASA 81mg
  Other Names: aspirin
  Arms: Len-Dex+ASA

SUMMARY:
The intended study is designed as a a phase IV pragmatic multicenter randomized controlled clinical trial, comparing the impact of two different therapies including ASA vs. Rivaroxaban in newly diagnosed or relapsed and refractory multiple myeloma patients treated with Lenalidomide Dexamethasone (Len-Dex) combination therapy. The pilot feasibility study was conducted in preparation for this randomized controlled trial designed to assess the effect of an intervention.

DETAILED DESCRIPTION:
RithMM is a phase IV, pragmatic, multicenter, open label Canadian trial. The study started with a pilot feasibility phase where 3 centres (London, Ottawa and Halifax) enrolled 34 patients within 12 months. Utilizing a roll-over design, the full RithMM trial will require a total of 304 patients to demonstrate that rivaroxaban 10 mg daily for 6 months is superior to ASA 81 mg daily for 6 months in preventing any thromboembolic events in newly diagnosed myeloma (NDMM) and relapsed/refractory (RRMM) patients on Len-Dex -based therapy. The study will require 8 participating centres in order to be able to achieve our recruitment goal within 12 to 18 months. Patients with NDMM or RRMM receiving Len-Dex based combination therapy with or without combination with other anti-myeloma drugs will be assessed for eligibility to be enrolled in the study. The research team intends to rollover the participants of our feasibility study into this current full randomized control trial comparing the efficacy outcome for the RithMM trial is the overall incidence of cardiovascular events, which includes arterial or venous thromboembolic events.

By conducting this trial, the investigators plan to externally validate the International Myeloma Working Group (IMWG) criteria model for thromboembolic risk by assessing the relevance of measuring pre-specified myeloma and thrombosis activity biomarkers (D-Dimer, beta-2 microglobulin, C-reactive protein (CRP), LDH) at every follow-up visit and their potential association with thromboembolism (TE) risk.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Multiple Myeloma
2. Scheduled to start on Len-Dex therapy
3. Be ≥ 18 years of age
4. Able to provide written informed consent
5. Pre-clinical laboratory must meet the following criteria at enrollment

   * Platelet count >50 × 109/L
   * Creatinine clearance (CrCl) >15mL/min using Cockcroft-Gault Equation

Exclusion Criteria:

1. Major bleeding event within the previous 3 months prior to commencement of Len Dex therapy
2. Documented severe liver disease in the past 6 months (eg. acute clinical hepatitis, chronic active hepatitis, or cirrhosis)
3. Patient with a history of antiphospholipid syndrome especially if he/she is triple positive for lupus anticoagulant, anticardiolipin antibodies, and/or anti-b2 glycoprotein I antibodies.
4. A history of malignancy (with the exception of MM) within 2 years before randomization or any previously diagnosed malignancy with evidence of residual disease. Patients with a history of basal cell or squamous carcinoma are not excluded.
5. Patient with history of gastric or duodenal ulcer within 2 years
6. Plasma cell leukemia; systemic amyloidosis
7. Patient on therapeutic anticoagulation for treatment of VTE or ATE, or stroke prevention in non-valvular atrial fibrillation. Patients with a previous history of VTE who are not on any active anticoagulant therapy will not be excluded.
8. Patient on antiplatelet agents due to an absolute indication (e.g.; coronary stent, carotid stent).
9. Patients receiving concomitant systemic treatment with strong inhibitors of both CYP3A4 and P-gp such as ketoconazole, itraconazole, posaconazole or ritonavir)
10. Patient on single agent lenalidomide
11. Life expectancy less than 3 months as determined by the investigator.
12. Unstable medical or psychological condition that would interfere with trial participation, as determined by the investigator
13. Patient not able or not willing to give consent to participate in the study
14. Uncontrolled cardiovascular disease within 6 months prior to enrollment
15. Uncontrolled or poorly controlled diabetes or renal disease
16. Major surgery within 2 weeks before randomization
17. Known allergies, hypersensitivity, or intolerance to any of the study drugs.
18. Patients not able or not willing to give consent to participate in the Study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of venous thromboembolic (VTE) and/or arterial thromboembolic (ATE) events in patients with Multiple Myeloma placed on the Rivaroxaban vs Aspirin after starting with Len-Dex therapy | 6 months
  At each visit, patients will be asked standardized questions to capture the presence of primary. During these interviews the study coordinator will collect data related to resource utilization (e.g. health care services use) and ask whether the patient had a diagnosis of VTE, ATE or a bleeding event during this period. Any hospital or medical office encounters associated to any of the above-mentioned complaints will be checked and any test or procedures done will be recorded (e.g; echocardiogram, ECG, CT scan, MRI, transfusion).
Number of participants with treatment-related adverse events as assessed by CTCAE v6.0 | 6 months
  Frequency and severity of adverse events and serious AEs based on hospital admission and patient-self reporting events

SECONDARY OUTCOMES:
External validation of the IMWG criteria for risk assessment of thromboembolic events in multiple myeloma patients | 6 months
  Subgroup analysis stratifying patients into low and high risk of thromboembolic events to assess any potential difference in the efficacy and safety outcomes.
Assessment of correlation of between levels of biomarkers of myeloma and thrombosis with the risk of ATE or VTE | 6 months
  The bio-markers are: D-dimer, LDH, B2 microglobulin and C-reactive protein (CRP) will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Martha Louzada, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamat AV Rivaroxaban Is an Effective and Well Tolerated Anti Thrombotic Agent in Patients on Lenalidomide Therapy and in Multiple Myeloma Blood 2014 124:5095;
- [Result] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Result] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Result] Palumbo A, Rajkumar SV, Dimopoulos MA, Richardson PG, San Miguel J, Barlogie B, Harousseau J, Zonder JA, Cavo M, Zangari M, Attal M, Belch A, Knop S, Joshua D, Sezer O, Ludwig H, Vesole D, Blade J, Kyle R, Westin J, Weber D, Bringhen S, Niesvizky R, Waage A, von Lilienfeld-Toal M, Lonial S, Morgan GJ, Orlowski RZ, Shimizu K, Anderson KC, Boccadoro M, Durie BG, Sonneveld P, Hussein MA; International Myeloma Working Group. Prevention of thalidomide- and lenalidomide-associated thrombosis in myeloma. Leukemia. 2008 Feb;22(2):414-23. doi: 10.1038/sj.leu.2405062. Epub 2007 Dec 20. PMID 18094721
- [Result] Al-Ani F, Bermejo JM, Mateos MV, Louzada M. Thromboprophylaxis in multiple myeloma patients treated with lenalidomide - A systematic review. Thromb Res. 2016 May;141:84-90. doi: 10.1016/j.thromres.2016.03.006. Epub 2016 Mar 5. PMID 26986753
- [Result] Levine MN, Gu C, Liebman HA, Escalante CP, Solymoss S, Deitchman D, Ramirez L, Julian J. A randomized phase II trial of apixaban for the prevention of thromboembolism in patients with metastatic cancer. J Thromb Haemost. 2012 May;10(5):807-14. doi: 10.1111/j.1538-7836.2012.04693.x. PMID 22409262
- [Result] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Result] Leleu X, Rodon P, Hulin C, Daley L, Dauriac C, Hacini M, Decaux O, Eisemann JC, Fitoussi O, Lioure B, Voillat L, Slama B, Al Jijakli A, Benramdane R, Chaleteix C, Costello R, Thyss A, Mathiot C, Boyle E, Maloisel F, Stoppa AM, Kolb B, Michallet M, Lamblin A, Natta P, Facon T, Elalamy I, Fermand JP, Moreau P. MELISSE, a large multicentric observational study to determine risk factors of venous thromboembolism in patients with multiple myeloma treated with immunomodulatory drugs. Thromb Haemost. 2013 Oct;110(4):844-51. doi: 10.1160/TH13-02-0140. Epub 2013 Aug 1. PMID 23903204
- [Derived] Kahale LA, Matar CF, Tsolakian I, Hakoum MB, Yosuico VE, Terrenato I, Sperati F, Barba M, Hicks LK, Schunemann H, Akl EA. Antithrombotic therapy for ambulatory patients with multiple myeloma receiving immunomodulatory agents. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD014739. doi: 10.1002/14651858.CD014739. PMID 34582035